CLINICAL TRIAL: NCT00984997
Title: Phase II Study of Combined Modality Treatment for Resectable Non-Small Cell Superior Sulcus Tumors
Brief Title: Combined Modality Treatment for Resectable Non-Small Cell Superior Sulcus Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID92-038
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: Superior Sulcus Tumor; Lung Cancer; Non-Small Cell; Multimodality Treatment; Surgery; Segmentectomy; Lobectomy; Cisplatin; CDDP; Etoposide; VP-16; VePesid; Radiation Therapy; Radiotherapy; Chest Irradiation; Prophylactic Cranial Irradiation; PCI
MeSH Terms: conditions — Lung Neoplasms; Pancoast Syndrome | interventions — Surgical Procedures, Operative; Radiotherapy; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery + Radiotherapy + Chemotherapy (Experimental): Surgery followed by radiotherapy and chemotherapy started at the beginning of radiotherapy. Segmentectomy or lobectomy with en bloc resection of the involved chest. Radiation therapy consists of 60 Gy in 50 fractions for negative margins, or 64.8 Gy in 54 fractions for positive margins, at 1.2 Gy per fraction, 2 fractions per day, 5 days per week. Cisplatin 50 mg/M^2 given intravenously on days 1 and 8; the cycle will be repeated beginning on day 29.
  Etoposide given by mouth 30-60 minutes prior to each administration of radiotherapy, on days 1-5 and days 8-12; the cycle will be repeated beginning day 29. Prophylactic Cranial Irradiation 25 Gy in 10 fractions of 2.5 Gy, 1 fraction per day, will be given at the completion of chest irradiation, and is optional.
  Interventions: Procedure: Surgery; Radiation: Chest Irradiation; Drug: Cisplatin; Drug: Etoposide; Radiation: Prophylactic Cranial Irradiation

INTERVENTIONS:
Procedure: Surgery — Segmentectomy or lobectomy with en bloc resection of the involved chest.
Radiation: Chest Irradiation — Radiation therapy consists of 60 Gy in 50 fractions for negative margins, or 64.8 Gy in 54 fractions for positive margins, at 1.2 Gy per fraction, 2 fractions per day, 5 days per week.
  Other Names: Radiotherapy
Drug: Cisplatin — 50 mg/M^2 given intravenously on days 1 and 8; the cycle will be repeated beginning on day 29.
  Other Names: Platinol; CDDP
Drug: Etoposide — given by mouth 30-60 minutes prior to each administration of radiotherapy, on days 1-5 and days 8-12; the cycle will be repeated beginning day 29.
  Other Names: VePesid; VP-16
Radiation: Prophylactic Cranial Irradiation — 25 Gy in 10 fractions of 2.5 Gy, 1 fraction per day, will be given at the completion of chest irradiation, and is optional.
  Other Names: PCI

SUMMARY:
1. To determine the outcome of patients with potentially resectable superior sulcus tumors of non-small cell histology treated by surgery followed by accelerated radiation therapy and chemotherapy.
2. To evaluate toxicity, the initial local-regional control rate, sites of and time to local and distant failures.

DETAILED DESCRIPTION:
Eligible (surgically resectable and medically operable) patients will have surgery followed by radiation therapy, given twice daily, for 5 weeks if margins are negative and for 5-1/2 weeks for positive margins. Grossly positive margins can be treated by brachytherapy followed by external radiotherapy.

Concomitant chemotherapy consisting of cisplatin given intravenously on days 1 and 8, and etoposide taken by mouth 30-60 minutes prior to each radiotherapy treatment x the first 10 days. The cycle will be repeated start day 29.

If the patients are considered to have no evidence of disease in one month after completion of chemotherapy, optional prophylactic radiotherapy to the brain will be give in 10 fractions once daily for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. No previous treatment.
2. Tumor must be resectable.
3. >/= 18 and </= 70 years of age.
4. Zubrod performance status </= or higher performance status if based only on pain.
5. Must have adequate bone marrow, liver and renal function as defined in 3.6.

Exclusion Criteria:

1. Cytological or histological proof of N3 disease.
2. Evidence of metastatic disease to distant sites.
3. Patients with impending cord compression will be ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1993-10; Primary Completion 2007-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rates of Locoregional control (LRC) [Response] Following Surgery and Accelerated Radiation Therapy/Chemotherapy | Assessed from one month after completion of chemotherapy to year 10
  Locoregional control (LRC) defined as disease non-recurrence in a localized area for patients with resectable superior sulcus tumors treated with surgical resection followed by adjuvant chemoradiation. LRC measured as percentage of participants without recurrence at rates of local control as measured Years 2, 5, and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Ritsuko Komaki, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org